CLINICAL TRIAL: NCT06803251
Title: Il Ruolo Del Chirurgo Vascolare Nella Chirurgia Oncologica Delle Masse Addominali E Pelviche Retroperitoneali
Brief Title: The Role of the Vascular Surgeon in Oncologic Surgery of Abdominal and Pelvic Retroperitoneal Masses
Acronym: IOVA-rpt
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IOVA-rpt
Record Dates: First submitted 2024-11-28; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Retroperitoneal Neoplasms
MeSH Terms: conditions — Retroperitoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retroperitoneal tumors (RPTs - retroperitoneal tumors) are neoplasms that originate from the soft tissues of the retroperitoneum and in their more invasive forms can involve the retroperitoneal organs and large abdominal and pelvic vascular structures. They are divided into benign tumors (20%), of which teratomas and tumors of neurogenic origin are the most frequent, and malignant tumors (80%), of which the most frequent are sarcomas (RPS - retroperitoneal sarcoma)1.

These are often large lesions, which can exceed 15 cm in diameter and which develop asymptomatically until the surrounding structures are involved. The initial symptoms are often represented by lumbar pain and abdominal distension which occur after multiple organ involvement.

To date, the treatment of choice is surgical excision of the mass with the aim of obtaining a clean resection margin R0 (macroscopically and microscopically free of disease) or R1 (with margin only macroscopically free of disease).

The most recent literature on this topic demonstrates how the treatment of RPS in specialized centers by a multidisciplinary team that works as a team and uses cutting-edge diagnostic and surgical techniques can improve the R0/R1 resection rate and overall survival. (OS)2.

The rate of intra- and post-operative surgical complications increases in direct proportion to the width of the excision; however, major complications are not associated with statistically significant differences in terms of OS, local recurrence (LR) and survival in the absence of distant metastases

DETAILED DESCRIPTION:
Very large abdominal and pelvic retroperitoneal masses frequently involve the retroperitoneal vascular structures.

Data from the literature show that after spinal surgery and orthopedic surgery, oncological surgery represents a specialist branch that frequently requires intraoperative vascular surgical assistance (6.7 - 9.6% of requests)5,6

. In these cases, the surgical assistance of the vascular surgeon allows the safe removal of the mass, the possible repair of the vessels damaged during cleavage and isolation of the mass, ligation or complete reconstruction of the vascular segment involved and contributes to reducing intraoperative and postoperative complications.

The clinical relevance of the evaluation of the short- and long-term results of the study lies in the fact that the case study it is expected to obtain greatly exceeds the few already published. Knowledge of outcomes on a larger sample will help shed light on aspects such as the need for more or less extensive surgical resection and on the choice of revascularization technique.

The primary objective of the study is to evaluate the outcomes of musculoskeletal tumor removal procedures in relation to the type of vascular surgical care provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a retroperitoneal mass involving the abdominal and/or pelvic vascular structures and requiring surgical removal
* Planned surgical treatment with intra-operative assistance from the vascular surgeon
* Obtaining informed consent
* Age 18 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belonging to the UU.OO. General Surgery, Urology and Gynecological Oncology of the IRCCS University Hospital of Bologna, with diagnosis of intra-abdominal or pelvic retroperitoneal mass with involvement of vascular structures and indication for surgical treatment of removal of the mass which requires the presence of a vascular surgeon. This indication is supported by international guidelines and represents normal clinical practice in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of vascular issues during the procedure | From the first patient enrolled to the 70th patient, an average of 3 years
  Numbers of major and minor vascular issues during retroperitoneal procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italia, Italy